CLINICAL TRIAL: NCT03625999
Title: A Novel Intervention for Training Auditory Attention in Adolescents With Autism Spectrum Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Our study stopped before it could begin because of the Covid-19 pandemic. We revised the study so that it could be performed virtually, but the revised study isn't a clinical trial.
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Helen B. Tager-Flusberg, Principal Investigator, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 4875E
Record Dates: First submitted 2018-08-06; First posted 2018-08-10 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Auditory attention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Parents and children selected for the Training group will be lent a laptop for the duration of the at-home training, and assisted in opening the video game training exercise. Parents and children will be shown the game's operation and controls, including a home visit to the family's house to help them establish the game as part of routine. Parents will be asked to engage their children in the video game training exercise (on the laptop) for a minimum of 20 minutes, 3 times a week, for 4 weeks. The app will log all responses as well as time spent playing.
  Interventions: Behavioral: video game training exercise
- Wait-List Control (No Intervention): The families assigned to the wait-list control group will not receive access to the game until after 4 weeks and completion of the secondary round of testing at the lab. After the second lab visit and completion of the testing, families will be given access to the video game training exercise (on a loaned laptop), walked through the game's operation and controls, and encouraged to use it as often as they or their child like. If the child plays the game for a minimum of 20 minutes, 3 times per week, for 4 weeks, the family will be invited back to CARE for post-testing.

INTERVENTIONS:
Behavioral: video game training exercise — The game, called "The Silent Service" and developed by our collaborators, is an online game with an underwater theme, and is comprised of 5 distinct mini-games, each of which demands auditory attention. The mission is to navigate an underwater scene, listening and responding to 'sonar' (e.g., an oddball in a stream of sounds). For example, participants may have to respond to an oddball sound stream to protect their submarine from a looming sea monster, while successfully ignoring a distractor sound stream (responses to the distractor sound stream allow the sea monster to damage the submarine). The five games share the same underlying framework of detecting oddballs while ignoring distractors but have unique artwork and 'backstories' to keep players interested. There is a hierarchical reward structure for 'leveling up' across the game that helps players to stay engaged and interested while playing.
  Other Names: game
  Arms: Training Group

SUMMARY:
Background: Previous research has shown that individuals with ASD often have difficulties coping with auditory stimuli in the environment. These difficulties can be extremely debilitating, lead to anxiety and disruptive behaviors, and interfere with the ability to process and understand speech.

Research Design: In previous research, the investigators have identified a brain marker associated with poor auditory attention that can provide a direct readout of auditory processing issues. The investigators will develop and test a cognitive/behavioral intervention (a tablet-based game app) that is highly engaging and accessible to a wide range of individuals with ASD. The intervention is designed to train adolescents with ASD to adapt and attend to auditory cues.

Objectives: To evaluate whether the intervention leads to improvement in auditory attention as assessed by behavior changes over the course of training; to investigate the impact of the intervention on behavioral assessment of problems hearing speech in noisy environments, neural processing of sounds, and changes in parent report on responses to sounds that impact that daily lives of the participants; and finally- to determine which adolescents with ASD benefit the most and least from interventions such as this one.

We hypothesize that we can elicit changes in the neural processing of sounds for adolescents with ASD via training in the form of the tablet-based game we are developing. If we are successful, this could lead to other interventions for persons with ASD in the hopes of improving the auditory difficulties they face.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent children and young adults, both males and females;
* Between the ages of 13:0 and 20:11 years of age
* Speak or hear English at home at least 50% of the time
* Meet criteria for a confirmed diagnosis of Autism Spectrum Disorder.

Exclusion Criteria:

* Nonverbal mental age below 18 months
* Insufficient manual dexterity that would prevent working with a tablet or phone-based app

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Child Behavioral Assessment: ADOS | 4-6 weeks
  All participants will come back to the center after 4 weeks to complete post-test behavioral assessments, including ADOS (Autism Diagnostic Observation Scale). The ADOS measures autism signs and symptoms. The minimum and maximums range depending on the specific module used (ADOS is available in many modules, the appropriate module to use is selected by the expressive language ability of the participant), but in general, higher scores on the ADOS indicate more severe or widespread symptoms.
Child Behavioral Assessment: Leiter-3 | 4-6 weeks
  All participants will come back to the center after 4 weeks to complete post-test behavioral assessments, including Leiter-3. The Leiter-3 is a nonverbal intelligence assessment, and measures attention, activity level, mood regulation, organizational skills, anxiety, sociability, impulse control, energy & feelings, and sensory reactivity. The range of composite scores is 30-170, and higher numbers indicate higher intelligence scores. The ranges encompass 'severe delay' to 'extremely high/gifted' so it can be used with persons of any ability.
Child Behavioral Assessment: PPVT-5 | 4-6 weeks
  All participants will come back to the center after 4 weeks to complete post-test behavioral assessments, including PPVT-4. The PPVT-4 (Peabody Picture Vocabulary Test) is a booklet containing pictures of commonly known items or objects, used to test receptive vocabulary, for example with verbal prompts such as "Which one is window?", or "Show me phone." The item is scored in terms of % correct responses, with a higher % correct indicating a bigger receptive vocabulary.
Child Behavioral Assessment: EVT-3 | 4-6 weeks
  All participants will come back to the center after 4 weeks to complete post-test behavioral assessments, including EVT-2. EVT-2 is a measure of expressive vocabulary and word retrieval. It can be used to quickly assess expressive vocabulary without requiring reading or writing. Standard scores range from 20 to 160, encompassing 'extremely low' to 'extremely high' so it can be used with persons of any english language ability. Higher scores indicate higher expressive language ability.
Parent Questionnaire: SCQ | 4-6 weeks
  All participants will come back to the center after 4 weeks to have parents or caregivers complete post-test behavioral questionnaires, including the SCQ (Social Communication Questionnaire). The SCQ was designed to evaluate communication skills and social functioning in children who may have ASD, and consists of yes-or-no questions so that it can be completed quickly. Higher scores indicate more severe or widespread symptoms.
Parent Questionnaire: VABS-3 | 4-6 weeks
  All participants will come back to the center after 4 weeks to have parents or caregivers complete post-test behavioral questionnaires, including the VABS-3 (Vineland Adaptive Behavior Scales). The Vineland provides scores for adaptive behavior domains (Communication, Daily Living Skills, Socialization, Motor Skills and Maladaptive Skills), and is designed to assess ability for self-sufficiency based on its ability to measure personal skills needed for everyday life. For each subdomain, scores range from 1 to 24, and for total scores, the range is 20 to 140. In both cases, higher scores indicate a positive ability to use or employ an adaptive behavior in place of a personal weakness or difficulty, so a better ability to work around one's limitations.
Parent Questionnaire: RBS-R | 4-6 weeks
  All participants will come back to the center after 4 weeks to have parents or caregivers complete post-test behavioral questionnaires, including the RBS-R (Repetitive Behavior Scales, revised). The RBS-R provides a quantitative, continuous measure of the full spectrum of repetitive behaviors, consisting of six subscales (Stereotyped behavior, Self-Injurious behavior, Compulsive behavior, Routine behavior, Sameness behavior, and Restricted behavior). Each behavior listed within each subscale is scored on a scale of 0 to 3, where 0 means a behavior does not occur and 3 means a behavior is a severe problem. As such, for the total score, a higher score means more extreme repetitive behaviors.
Parent Questionnaire: SSP | 4-6 weeks
  All participants will come back to the center after 4 weeks to have parents or caregivers complete post-test behavioral questionnaires, including the SSP (Short Sensory Profile). The sensory profile is a measure of responses to sensory events in daily life. There are several sections, encompassing a range of sensory experiences (tactile, taste/smell, movement, seeks sensation, auditory filtering, low energy/weak, and visual/auditory sensitivity), and the total score ranges between 38 and 190, with 38 and other low numbers reflecting an extreme difference from typically developing peers, and 190 and other high numbers reflecting a similarity to typically developing peers.
Parent Questionnaire: CASI-5 | 4-6 weeks
  All participants will come back to the center after 4 weeks to have parents or caregivers complete post-test behavioral questionnaires, including the CASI-5 (Child and Adolescent Symptom Inventory). The CASI-5 is a behavior rating scale that assesses symptoms of a range of 15 different developmental, emotional, and behavioral disorders that can be used to assess any comorbidities a subject may display symptoms for. The scores (total range 0-100) are calculated depending on several factors, but in general, higher numbers indicate the presence of more symptoms (of any disorder) and lower numbers indicate fewer symptoms or less impairment.
Post-test EEG | 4-6 weeks
  All participants will come back to the center after 4 weeks to complete post-test EEG testing. Participants will wear an EEG net connected with elastic threads while listening to sound series designed to assess attention to distinctive sounds. During the task, investigators will assess waveforms alpha, beta, theta, gamma and delta to look for differences in auditory processing between first visit and post-test visit.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Tager-Flusberg, PhD, Study Chair — Prinicipal Investigator
Locations (1):
- Center for Autism Research Excellence, Boston, Massachusetts, United States